CLINICAL TRIAL: NCT06599944
Title: The Role of Contact in Nursing Students' Attitudes Towards Immigrant Individuals and Cultural Intelligence: a Comparative Study
Brief Title: Contact and Attitudes in Nursing Students: Immigrants and Cultural Intelligence
Status: Enrolling by invitation | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Aytuğ Türk, RN, PhD, Research Assistant, Muğla Sıtkı Koçman University
Other Study IDs: MSKU-SBF-AT-01
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Being a Third-year Nursing Student At the Faculty of Nursing, Ege University During the 2023-2024 Academic Year; Having Completed a Nursing Practice At a Migrant Health Center
Keywords: Cultural Intelligence; Nursing Students; Immigrant Attitudes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Students who applied Diseases and Nursing Care 3 at the Migrant Health Centre: Students who carry out the application for the Diseases and Nursing Care 3 course at the Migrant Health Centre will be included in this group and the relevant measurement tools will be applied.
  Interventions: Diagnostic Test: Negative Attitude Scale towards Immigrant Individuals and Cultural Intelligence Scale
- Students who practiced Diseases and Nursing Care 3 in a unit other than the Migrant Health Centre: Related measurement tools will be applied to students who perform the practice for the Diseases and Nursing Care 3 course in a different unit other than the migrant health centre.
  Interventions: Diagnostic Test: Negative Attitude Scale towards Immigrant Individuals and Cultural Intelligence Scale

INTERVENTIONS:
Diagnostic Test: Negative Attitude Scale towards Immigrant Individuals and Cultural Intelligence Scale — Negative Attitude towards Immigrant Individual and Cultural Intelligence scales will be applied to the students in both groups included in the study. Thus, to measure the change in negative attitudes towards immigrant individuals and cultural intelligence as a result of the practice in the migrant health centre.

SUMMARY:
The study aims to determine the effect of practice in a migrant health center on students' intercultural sensitivity and ethnocentrism. In this context, it is planned to be conducted between December 2022 and February 2023 as a causal-comparative study with students who have completed the Diseases and Nursing Care 3 course at the Faculty of Nursing, Ege University.

The research group will consist of 50 students who completed the Diseases and Nursing Care 3 course practice at the Migrant Health Center during the 2021-2022 academic year. The comparison group will consist of 50 students who completed the same course practice in a different unit, selected through simple random sampling (random selection of student names placed in a bag). The 'Personal Information Form,' 'Cultural Sensitivity Scale,' and 'Ethnocentrism Scale' will be used as data collection tools. The data obtained will be analyzed using SPSS (Statistical Package for Social Sciences) for Windows 22.0 software.

DETAILED DESCRIPTION:
Migration is a population movement in which people relocate individually or collectively, regardless of the cause, structure, or duration. These movements can be voluntary or forced, driven by natural disasters, armed conflicts, or political and economic reasons. According to the Glossary of Migration Terms, a migrant is someone who moves to a different country or region to improve the material and social conditions of themselves and their family, and to enhance their life expectations, without being influenced by coercive external factors.

The Syrian Civil War led to the migration of more than five million Syrians to Turkey, Lebanon, Jordan, and other countries. In Turkey alone, there are 3.6 million Syrian migrants. This influx has highlighted the need to develop migration and migrant health policies for Syrian migrants in the country. Although Syrian migrants have been in Turkey for an extended period, they face significant challenges, particularly due to the language barrier, which hinders their ability to express themselves and communicate effectively. While some communication is possible in border provinces where there are shared cultural and linguistic characteristics, difficulties increase as migrants move towards the western regions of the country.

Migrants in Turkey face challenges in various areas, including accommodation, education, employment, and access to health services, in addition to language barriers. To address these issues, Migrant Health Centres (MHCs) were established as part of the SIHHAT project. The Ministry of Health has been setting up MHCs across the country since 2015. These centers provide free primary healthcare services to unregistered migrants without temporary protection identity documents and non-Syrian migrants. MHCs are designed to offer primary health care services to migrants under temporary protection in Turkey, with one unit serving every 4,000 people, in line with the standards of family medicine in the country. By employing Turkish and Syrian healthcare personnel and Arabic- and Turkish-speaking patient guidance personnel, these centers aim to overcome the challenges posed by language and cultural barriers and deliver effective healthcare services.

In Turkey, the formation of multicultural societies due to migration, driven initially by war and later by economic, political, and sociological factors, has impacted the provision of services, including healthcare. This has underscored the importance of intercultural sensitivity. Intercultural care plays a crucial role in nursing. Nursing philosophy emphasizes the necessity of providing individual-centered care to all ethnic groups in a globalizing world. Leininger's Cultural Care Theory highlights the importance of nurses developing their knowledge and skills related to cultural differences and being aware of their patients' values, beliefs, and lifestyles. Nursing practices involve providing holistic care to patients, which requires cultural competence and consideration of cultural differences. Nurses develop intercultural sensitivity when they acknowledge that the individuals they care for are culturally different from themselves and when they respect and appreciate these cultural characteristics.

Although providing individual-centered intercultural care is a nurse's responsibility, there are instances where nurses may exhibit ethnocentric attitudes due to a lack of knowledge, understanding, awareness, education, cultural competence, or beliefs about culture. Ethnocentrism, defined as the belief in the superiority of one's own culture and the tendency to judge other cultures by one's own cultural values, can lead to patient alienation, inadequate treatment, misdiagnosis, and culturally inappropriate healthcare services. However, a culturally sensitive approach can improve the quality of care, increase patient satisfaction, enhance health outcomes, and reduce stress and burnout. In this context, acquiring intercultural sensitivity also implies a reduction in ethnocentrism. Nurses, as healthcare professionals, are responsible for providing care to individuals with diverse cultural backgrounds. Therefore, it is essential to assess the levels of intercultural sensitivity and ethnocentrism during their training period to enhance the cultural competence of future nurses. It is believed that the levels of cultural sensitivity and ethnocentrism among nursing students working with migrants in MHCs are shaped through direct contact and interaction with migrant individuals during their practical training.

ELIGIBILITY:
Inclusion Criteria:

* To be a 4th year student of Ege University Faculty of Nursing
* To have carried out the application for Diseases and Nursing Care 3 course.
* Accepting to participate in the research

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study, it was aimed to compare the intercultural sensitivity and ethnocentrism levels of nursing students who practice in migrant health centres and provide care to individuals from different cultures and nursing students who do not practice in migrant health centres.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
Negative Attitude Scale towards Immigrant Individuals Scale | 20.10.2024-01.11.2024
  The Negative Attitude towards Immigrant Individuals scale will be administered to students in both groups included in the study. The aim is to determine whether the practice at the migrant health center results in a difference in negative attitudes towards immigrant individuals. High scores on the scale indicate a higher level of negative attitudes towards immigrants.
Cultural Intelligence Scale | 20.10.2024-01.11.2024
  The Cultural Intelligence scale will be administered to students in both groups included in the study. The aim is to determine whether the practice at the migrant health center leads to differences in cultural intelligence. High scores on the scale indicate that the participants' cultural intelligence has been positively impacted and has increased.

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla Sıtkı Koçman University, Muğla, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 01.12.2024-31.12.2025
Access Criteria: All researchers who work as a researcher at a university and have an edu-linked e-mail address